CLINICAL TRIAL: NCT05585567
Title: A Single Center, Randomized, Open-labeled, Exploratory Clinical Study to Evaluate the Safety and Immunogenicity of Bivalent Vaccine V-01-B5 as a Booster Dose in Participants Aged 18-59 Years Vaccinated 3-dose Inactivated COVID-19 Vaccine
Brief Title: A Preliminary Exploratory Study to Evaluate the Safety and Immunogenicity of Omicron Variant Bivalent Vaccine V-01-B5
Acronym: COVID-19
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: V-01-B5- Booster-01
Record Dates: First submitted 2022-10-13; First posted 2022-10-19 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- V-01/V-01-B5 group (Experimental): One dose of V-01/V-01-B5
  Interventions: Biological: V-01/V-01-B5
- V-01-351/V-01-B5 group (Experimental): One dose of V-01-351/V-01-B5
  Interventions: Biological: V-01-351/V-01-B5
- V-01 group (Experimental): One dose of V-01
  Interventions: Biological: V-01

INTERVENTIONS:
Biological: V-01/V-01-B5 — Contains 10μg of V-01 and 10μg of V-01-B5
  Arms: V-01/V-01-B5 group
Biological: V-01-351/V-01-B5 — Contains 10μg of V-01-351 and 10μg of V-01-B5
  Arms: V-01-351/V-01-B5 group
Biological: V-01 — Contains 10μg of V-01
  Arms: V-01 group

SUMMARY:
It is a single center, randomized, open-labeled, exploratory clinical study to evaluate the safety and immunogenicity of Recombinant SARS-CoV-2 Fusion Protein bivalent Vaccine V-01-B5 as a second booster in adults aged 18-59 years after vaccinated with 3-dose of inactivated vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 -59 years old at time of consent, male or female;
* Normal body temperature;
* Participants who have completed 3-dose regimen of inactive vaccination (CoronaVac) against SARS-CoV-2 wild type in the past 5-9 months;
* Female participants who are not pregnant at the time of enrollment (urine pregnancy test is negative), nor during lactating; and has no birth plan and agree to take effective contraception in 7 months after enrollment; and took effective and acceptable contraceptive methods in the previous 2 weeks before the enrollment;
* Be able and willing to complete the study during the entire study and follow-up period;
* Participants who have the ability to understand the study process, sign the informed consent form voluntarily , and be able to comply with the requirements of the clinical study protocol.

Exclusion Criteria:

* Serious chronic diseases or uncontrolled diseases;
* Uncontrolled neurological disorders, epilepsy;
* Received any inactivated vaccine within 1 week or received any attenuated vaccines within 4 weeks;
* Patients with congenital or acquired immunodeficiency;
* History of severe allergy or be allergic to any components of the test vaccines;
* History of hereditary hemorrhagic tendency or coagulation dysfunction;
* Patients with malignant tumors and other patients have a life expectancy less than 1 year;
* Refuse to sign the informed consent form or inability to complete follow-ups as required by the protocol;
* History of previous COVID-19 infection;
* Pregnant or breastfeeding women, or females of childbearing potential who not agree to or able to take effective and acceptable contraceptive methods during the study;
* Participants who have participated in other clinical trials within 3 months or are participating in other clinical trials;
* Those considered by the investigator as inappropriate to participate in the study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2023-09-11 (Estimated)

PRIMARY OUTCOMES:
Adverse Event (AE) | 30 minutes after vaccination
  Observe the AEs occurs at different time point after vaccination
AEs | 0-7 days after vaccination
  Observe the AEs occurs at different time point after vaccination
AEs | 0-28 days after vaccination
  Observe the AEs occurs at different time point after vaccination
Serious adverse event (SAE) and adverse event of special interest (AESI) | Within 12 months after vaccination
  Observe the SAE and AESI after vaccination
Neutralizing antibody geometric mean titer (GMT) of Omicron BA.5 | 28 days after vaccination
  Neutralizing antibody GMT of the most prevalent SARS-CoV-2 variant (Omicron BA.5)

SECONDARY OUTCOMES:
Neutralizing antibody GMT of other SARS-CoV-2 variants | Until 12 months after vaccination
  Neutralizing antibody GMT of Delta variant and Omicron variants (BA.2, BA.4, BA.5)
Neutralizing antibody titer of other SARS-CoV-2 variants (MRNT) | Until 12 months after vaccination
  Neutralizing antibody titer of Delta variant and Omicron variants (BA.2, BA.4, BA.5) by MRNT
Neutralizing antibody titer of other SARS-CoV-2 variants (SVNT) | Until 12 months after vaccination
  Neutralizing antibody titer of Delta variant and Omicron variants (BA.2, BA.4, BA.5) by SVNT
Anti-SARS-CoV-2 receptor-binding domain (RBD) antibody level | Until 12 months after vaccination
  Anti-SARS-CoV-2 RBD antibody level after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Shaoguan Hospital of Chinese Medicine, Shaoguan, Guangdong, China